CLINICAL TRIAL: NCT06107881
Title: Beacon Sensors and Telerehabilitation to Assess and Improve Use of Devices (BeST-AID) for Low Vision
Acronym: BeST-AID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Nebraska (Other); New England College of Optometry (Other); Southern California College of Optometry at Marshall B. Ketchum University (Other); Mid-Michigan Eye Care (Unknown)
Responsible Party: Principal Investigator, Ava K. Bittner, OD, PhD, Associate Professor of Ophthalmology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BeST-AID 2.0
Record Dates: First submitted 2023-10-18; First posted 2023-10-30 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Low Vision; Low Vision Aids
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Intervention Model Description: randomized controlled non-inferiority trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telerehabilitation with low vision provider (Experimental): Low Vision Rehabilitation for use of magnification or visual assistive devices using videoconferencing for remotely delivered follow-up care
  Interventions: Behavioral: Low Vision Rehabilitation
- Usual Care In-Office (Active Comparator): Low Vision Rehabilitation in-office for use of magnification or visual assistive devices
  Interventions: Behavioral: Low Vision Rehabilitation

INTERVENTIONS:
Behavioral: Low Vision Rehabilitation — Evaluation and training with magnification or visual assistive devices for visually-impaired adults

SUMMARY:
One goal of this research is to conduct a non-inferiority trial of telerehabilitation versus in-office care to provide follow-up training to individuals with low vision to enhance their quality of life by using magnification devices and/or visual assistive mobile apps for important daily activities, such as reading and/or other valued tasks. This is a high priority given the increasing prevalence of low vision, paucity of low vision rehabilitation providers, and barriers related to access to care, such as transportation and geography, which can be essentially eliminated with telerehabilitation. Another goal of this project is to determine whether significant changes in environmental data collected by Bluetooth low energy beacon sensors can be used as a solution to monitor and indicate when low vision patients' have abandoned the use of their magnification devices, which has the potential to substantially enhance patient management by providing timely low vision rehabilitation services.

ELIGIBILITY:
Inclusion Criteria:

* adults with any level of vision loss due to any ocular disease who are age 18 and older, and who have received new magnification device(s) for the first time (i.e., hand-held optical magnifiers, portable electronic video magnifiers, high near add powers of +4.00 or greater, visual assistive mobile apps for their smartphone/tablet, some stand magnifiers and CCTVs) from one of our participating low vision rehabilitation sites at the four academic centers and one private practice.

Exclusion Criteria:

* schedules not permitting participation in planned study visits (including planning to move far from their clinical provider's office within the first 4-months of the study (i.e., cannot attend in-office visits) or take extended vacation that would not allow them to complete study procedures during the first four months of the study period),
* inability to understand study procedures or communicate responses to visual stimuli in a consistent manner (greater than mild cognitive impairment as per TICS),
* substance abuse,
* significant hearing loss (unable to hear communication by phone or via videoconferencing),
* significant medical condition likely to limit participation or lifespan,
* individuals who require other types of LVR training or intervention (e.g., psychosocial).
* For Bluetooth low energy beacon sensors, exclusion would occur if their magnifier device has features that would not work in conjunction with the beacon sensors: (1) hands-free and do not have a place where the patient's hand is holding the device during use (therefore, they would not register a significant change in temperature), (2) no surface area of at least 1"x1" to which the beacon sensor could be attached without interfering with the device, or (3) use of visual assistive mobile apps only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Activity Inventory | changes from 1 month to 4 months to 8 months to 12 months to 13 months after receiving a magnification device
  questionnaire; scores will be Rasch analyzed in logic units with higher or positive scores indicating less difficulty (i.e., improvement)

SECONDARY OUTCOMES:
MNread | baseline, 1 month, 4 months, 8 months, 12 months, 13 months
  reading speed and acuity test
Sustained Silent Reading Test | baseline, 1 month, 4 months, 8 months, 12 months, 13 months
  prolonged reading test
International Reading Speed Text (IReST) | baseline, 1 month, 4 months, 8 months, 12 months, 13 months
  reading speed test
Radner Reading Charts | baseline, 1 month, 4 months, 8 months, 12 months, 13 months
  reading speed and acuity test
Vision rehabilitation satisfaction survey | after each session that will occur over a period of 1 to 8 months and and again at about 1 year
  surveys: post-telerehabilitation or in-office visits
Informant surveys by close acquaintances of participants | 4 months, 8 months, 12 months, 13 months
  survey
Adherence to hand-held optical magnifier use (frequency and duration) | baseline to 13 months
  Bluetooth low energy beacon sensor data

CONTACTS AND LOCATIONS:
Overall Officials: Ava K Bittner, OD, PhD, Principal Investigator — University of California, Los Angeles
Locations (9):
- United States (9):
  - Southern Califonia College of Optometry, Fullerton, California
  - Chan Family Optometry, Grass Valley, California
  - UCLA Stein Eye Institute, Los Angeles, California
  - Frank Stein & Paul S. May Center for Low Vision Rehabilitation at The Eye Institute, San Francisco, California
  - See What You Miss Optometry, Santa Monica, California
  - New England College of Optometry, Boston, Massachusetts
  - Boston University Eye Associates, Inc., Brockton, Massachusetts
  - Mid-Michigan Eye Care, Midland, Michigan
  - University of Nebraska: Weigel Williamson Center for Visual Rehabilitation at the Truhlsen Eye Institute, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: Undecided
Please contact the principal investigator

REFERENCES:
- [Background] Kaminski JE, Yoshinaga PD, Chun MW, Yu M, Shepherd JD, Chan TL, Deemer A, Bittner AK; BeST-AID Study Team. Value of Handheld Optical Illuminated Magnifiers for Sustained Silent Reading by Visually Impaired Adults. Optom Vis Sci. 2023 May 1;100(5):312-318. doi: 10.1097/OPX.0000000000002013. Epub 2023 Mar 22. PMID 36951854
- [Background] Bittner AK, Yoshinaga PD, Rittiphairoj T, Li T. Telerehabilitation for people with low vision. Cochrane Database Syst Rev. 2023 Jan 13;1(1):CD011019. doi: 10.1002/14651858.CD011019.pub4. PMID 36637057
- [Background] Bittner AK, Kaminski JE, Ross NC, Shepherd JD, Thoene SJ, Bui SZ, Yoshinaga PD; BeST-AID Study Team. Telerehabilitation Training to Facilitate Improved Reading Ability with New Magnification Devices for Low Vision. Optom Vis Sci. 2022 Oct 1;99(10):743-749. doi: 10.1097/OPX.0000000000001944. Epub 2022 Sep 6. PMID 36067410
- [Background] Bittner AK, Yoshinaga PD, Shepherd JD, Kaminski JE, Malkin AG, Chun MW, Chan TL, Deemer AD, Ross NC; BeST-AID Study Team. Acceptability of Telerehabilitation for Magnification Devices for the Visually Impaired Using Various Approaches to Facilitate Accessibility. Transl Vis Sci Technol. 2022 Aug 1;11(8):4. doi: 10.1167/tvst.11.8.4. PMID 35917136
- [Background] Malkin AG, Ross NC, Chun MW, Bittner AK; CARE Study Team. Why Are Visual Assistive Mobile Applications Underused by Low Vision Patients? Optom Vis Sci. 2022 Apr 1;99(4):333-334. doi: 10.1097/OPX.0000000000001893. No abstract available. PMID 35213868
- [Background] Bittner AK, Estabrook M, Dennis N. Bluetooth Low Energy Beacon Sensors to Document Handheld Magnifier Use at Home by People with Low Vision. Sensors (Basel). 2021 Oct 25;21(21):7065. doi: 10.3390/s21217065. PMID 34770374
- [Background] Bittner AK, Yoshinaga P, Bowers A, Shepherd JD, Succar T, Ross NC. Feasibility of Telerehabilitation for Low Vision: Satisfaction Ratings by Providers and Patients. Optom Vis Sci. 2018 Sep;95(9):865-872. doi: 10.1097/OPX.0000000000001260. PMID 30169361
- [Background] Bittner AK, Jacobson AJ, Khan R. Feasibility of Using Bluetooth Low Energy Beacon Sensors to Detect Magnifier Usage by Low Vision Patients. Optom Vis Sci. 2018 Sep;95(9):844-851. doi: 10.1097/OPX.0000000000001266. PMID 30169359